CLINICAL TRIAL: NCT03866005
Title: Prospective Study of Adjunctive Carotenoids Plus Anti-oxidants in Anti-VEGF Treated Diabetic Macular Edema
Acronym: PROACTIVEDME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ZeaVision, LLC (Industry)
Collaborators: Sound Retina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PROACTIVE-DME
Record Dates: First submitted 2019-03-05; First posted 2019-03-07 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Center-involved Diabetic Macular Edema (CI-DME)
Keywords: diabetes, retina, diabetic retinopathy, diabetic macular edema, anti-VEGF therapy
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy

STUDY DESIGN:
Intervention Model Description: This will be an investigator initiated, single-clinic/two location, double-blinded prospective study of 150 adult subjects with newly diagnosed CI-DME receiving anti-VEGF injections, with add-on laser and/or steroid as required on follow-up examination (Standard Treatment) versus standard treatment plus adjunctive DiVFuSS supplementation in one of two doses (2 softgels per day - Supplement Treatment Group 1; and 4 softgels per day - Supplement Treatment Group 2). Subjects will be identified and enrolled with informed consent from two retinal specialty practice sites in Washington State (Sound Retina; Tacoma, WA and Olympia, WA). Subjects will be randomized to Standard Treatment; Supplement Treatment Group 1, or Supplement Treatment Group 2.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: After enrollment by the study Primary Investigator, a single retinal specialist from each site, masked to subjects' supplement status, will deliver all treatments per his/her usual protocol for treatment of CI-DME based on individual examination findings. Supplements and identically-appearing placebo will be provided by ZeaVision, LLC of Chesterfield, MO.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo Arm - Standard Treatment (Placebo Comparator): 50 subjects with center-involved diabetic macular edema (CI-DME) and scheduled for treatment with intravitreal injection of anti-VEGF agents will receive softgel placebo containing canola oil, 2 capsules per day during the study duration
  Interventions: Other: canola oil placebo softgels, 2 per day
- Experimental Arm - 2 DiVFuSS formula softgel capsules (Experimental): 50 subjects receiving two DiVFuSS softgels per day
  Interventions: Dietary Supplement: Diabetes Visual Function Study (DiVFuSS) softgels
- Experimental Arm - 4 DiVFuSS formula softgel capsules (Experimental): 50 subjects receiving 4 DiVFuss softgels per day
  Interventions: Dietary Supplement: Diabetes Visual Function Study (DiVFuSS) softgels

INTERVENTIONS:
Dietary Supplement: Diabetes Visual Function Study (DiVFuSS) softgels — The adjunctive nutritional supplement will be the multi-component formula used in the Diabetes Visual Function Supplement Study (Western IRB number 1129944 Olympia, WA), containing the macular carotenoids lutein and zeaxanthin, as well as antioxidants (vitamins B1, B12, C, D, E, lipoic acid, coenzyme Q10, resveratrol), omega3 fatty acids (EPA/DHA) and botanical extracts (Pycnogenol™ [patented extract of French maritime pine bark, Pinus pinaster], grape seed and green tea extracts, curcumin).
  Arms: Experimental Arm - 2 DiVFuSS formula softgel capsules; Experimental Arm - 4 DiVFuSS formula softgel capsules
Other: canola oil placebo softgels, 2 per day — Placebo containing canola oil, 2 softgels per day
  Arms: Placebo Arm - Standard Treatment

SUMMARY:
This study will evaluate the effects of add-on carotenoid plus anti-oxidant nutritional supplementation to standard anti-vascular endothelial growth factor therapy for subjects with center-involved diabetic macular edema

DETAILED DESCRIPTION:
Diabetic retinopathy (DR) remains the leading cause of blindness in Americans of working age, and the majority of people with diabetes are expected to develop retinopathy, with as many as 10% developing sight-threatening retinopathy (proliferative retinopathy and/or center-involved macular edema) during their lifetime. Established risk factors for DR and diabetic macular edema (DME) include duration of disease, metabolic control (particularly severity and duration of hyperglycemia and hypertension), early age of diabetes diagnosis, male gender, Black and Hispanic race/ethnicity, and albuminuria (kidney disease). , In particular, DME accounts for the majority of vision loss due to diabetes, with significant impacts on activities of daily living and quality of life. Approximately 30% of patients with diabetes develop DME within twenty years of diagnosis.

Available treatments for DME include laser photocoagulation, intravitreal steroids via injection or sustained release implant and, most importantly, intravitreal injection of inhibitors of vascular endothelial growth factor (anti-VEGF). In a number of clinical trials, serial injections of anti-VEGF agents have demonstrated superiority for both reducing intra-retinal edema and improving/stabilizing visual acuity in patients with DME, and their use has become the recognized standard of care, particularly when DME is at or very near the foveal center (center-involved diabetic macular edema, CI-DME). However, anti-VEGF drugs for DME typically require multiple injections, are expensive, carry small but measurable risk of ocular and potentially systemic complications, and are not universally or adequately effective.

A number of biochemical processes have been elucidated as contributing factors in DME, including disruption of the cellular electron transport chain leading to excess production of mitochondrial reactive oxygen and nitrogen species (ROS and RNS) that drives accumulation of injurious glucose metabolites, with concomitant elevation of inflammatory cytokines, leukostasis, apoptosis (programmed cell death), retinal capillary leakage and release of vasoproliferative factors. More recent evidence has suggested that nutritional supplements may interfere with the pathogenesis of structural and functional abnormalities associated with diabetes and diabetic retinopathy. Specifically, use of a novel, multi-component, orally administered nutritional supplement was shown to improve visual function (contrast sensitivity, color perception, visual field) and serum markers of inflammation (hsCRP) in patients with non-proliferative diabetic retinopathy without affecting blood glucose control in an IRB-approved (Western IRB number 1129944 Olympia, WA) randomized, placebo-controlled clinical trial (The Diabetes Visual Function Supplement Study [DiVFuSS]

Hypothesis

Our aim is to test the hypothesis that adjunctive supplementation with the DiVFuSS formula, in addition to conventional anti-VEGF therapy with add-on laser photocoagulation and/or intravitreal steroid as necessary, will result in reduced macular edema, fewer required anti-VEGF injections and better visual acuity in treatment-naïve CI-DME subjects receiving therapy over two years in a retinal specialty clinic. A secondary outcome to be assessed is the percentage of patients requiring add-on laser or steroid treatment over the two years in each of the study groups.

Overview of Study Design

This will be an investigator initiated, single-clinic/two location, double-blinded prospective study of 150 adult subjects with newly diagnosed CI-DME receiving anti-VEGF injections, with add-on laser and/or steroid as required on follow-up examination (Standard Treatment) versus standard treatment plus adjunctive DiVFuSS supplementation in one of two doses (2 softgels per day - Supplement Treatment Group 1; and 4 softgels per day - Supplement Treatment Group 2). Subjects will be identified and enrolled with informed consent from two retinal specialty practice sites in Washington State (Sound Retina; Tacoma, WA and Olympia, WA). Subjects will be randomized to Standard Treatment; Supplement Treatment Group 1, or Supplement Treatment Group 2.

Study Allocation: 150 treatment-naïve subjects with CI-DME Requiring anti-VEGF therapy

Standard Treatment Group (50 participants) with treatment-naive center-involved diabetic macular edema will receive anti-VEGF therapy per specialists' usual protocol, with add-on laser or steroid if necessary (at specialist's discretion); Supplement Treatment Group 1 (50 participants) with treatment-naive center-involved diabetic macular edema will receive Standard Treatment plus two DiVFuSS softgels/day; Supplement Treatment Group 2 (50 participants) with treatment-naive center-involved diabetic macular edema will receive Standard Treatment plus four DiVFuSS softgels/day.

After enrollment by the study Primary Investigator, a single retinal specialist from each site, masked to subjects' supplement status, will deliver all treatments per his/her usual protocol for treatment of CI-DME based on individual examination findings. Supplements will be provided by ZeaVision, LLC of Chesterfield, MO. Subjects will receive detailed, dilated eye examinations with additional customary tests (measurement of visual acuity, spectral domain optical coherence tomography, high-resolution retinal photography) performed and recorded by the masked Primary Investigator at baseline, 3 months, 6 months,12 months, 18 months and 24 months. Follow-up phone calls will be performed monthly between visits to help assure compliance for the Test Supplement Treatment Groups (1 and 2). Wide-field fluorescein angiography (FA) will be performed at baseline, 12 months and 24 months per usual care and results recorded by the Primary Investigator.

Test Supplements

The adjunctive nutritional supplement will be the multi-component formula used in the Diabetes Visual Function Supplement Study (Western IRB number 1129944 Olympia, WA), containing the macular carotenoids lutein and zeaxanthin, as well as antioxidants (vitamins B1, B12, C, D, E, lipoic acid, coenzyme Q10, resveratrol), omega3 fatty acids (EPA/DHA) and botanical extracts (Pycnogenol™ [patented extract of French maritime pine bark, Pinus pinaster], grape seed and green tea extracts, curcumin).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed diabetes mellitus and treatment-naïve CI-DME requiring anti-VEGF therapy per retinal specialist's customary treatment regimen will be recruited to participate in the study. CI-DME will be defined as a central subfield thickness (CST) > 300 microns on spectral domain optical coherence tomography (SD-OCT) or CST > 250 microns with definite intra-retinal cystic fluid accumulation. Additional inclusion criteria are age > 18 years, and ability to give informed consent.

Exclusion Criteria:

* Age < 18 years, inability to give informed consent, evidence of proliferative diabetic retinopathy, evidence of other serious ocular disease (age-related macular degeneration, glaucoma, significant media opacity), history of previous intraocular surgery, including macular or panretinal photocoagulation (except uncomplicated cataract or keratorefractive surgery more than 6 months prior to enrollment), pregnant and nursing women, known sensitivity to any of the supplement ingredients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Best-corrected visual acuity | two years
  Best-corrected visual acuity at entry and conclusion of study
SD-OCT macular subfield thicknesses | two years
  Change in macular subfield thicknesses from baseline to study conclusion
Required number of anti-VEGF injections | two years
  The number of intravitreal anti-VEGDF injections required for treatment of center-involved diabetic macular edema

SECONDARY OUTCOMES:
Need for adjunctive laser photocoagulation and/or use of intravitreal steroids | two years
  The number of subjects in each arm requiring adjunctive laser photocoagulation or intravitreal steroids for treatment of CI-DME

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Sound Retina, Olympia, Washington
  - Sound Retina, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chous AP, Richer SP, Gerson JD, Kowluru RA. The Diabetes Visual Function Supplement Study (DiVFuSS). Br J Ophthalmol. 2016 Feb;100(2):227-34. doi: 10.1136/bjophthalmol-2014-306534. Epub 2015 Jun 18. PMID 26089210